CLINICAL TRIAL: NCT03244644
Title: A Phase 3 Prospective, Randomized, Double-blinded, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of RBX2660 (Microbiota Suspension) for the Prevention of Clostridium Difficile Infection
Brief Title: Microbiota Restoration Therapy for Recurrent Clostridium Difficile Infection (PUNCHCD3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-01
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Clostridium Difficile Infection (CDI)
Keywords: C Difficile Colitis; Clostridium Difficile; CDI; C.Difficile Diarrhea; Fecal Transplant; Fecal Microbiota Transplant (FMT); Microbiota Restoration Therapy; Diarrhea; FMT; Microbial Suspension
MeSH Terms: conditions — Clostridium Infections; Enterocolitis, Pseudomembranous; Diarrhea | interventions — Saline Solution; Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is an suspension of normal saline. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding
  Interventions: Drug: Placebo; Drug: Open label RBX2660 (only for confirmed CDI recurrence)
- RBX2660 (Experimental): RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation United States Pharmacopeia (USP) solution and cryoprotectant
  Interventions: Drug: RBX2660; Drug: Open label RBX2660 (only for confirmed CDI recurrence)

INTERVENTIONS:
Drug: RBX2660 — RBX2660 is a rectally administered microbiota suspension
  Other Names: microbiota suspension
  Arms: RBX2660
Drug: Placebo — Placebo is normal saline solution administered rectally
  Other Names: saline solution
  Arms: Placebo
Drug: Open label RBX2660 (only for confirmed CDI recurrence) — RBX2660 administered as a second treatment after confirmed CDI recurrence following the initial dose of placebo or RBX2660
  Other Names: microbiota suspension

SUMMARY:
This is a prospective, multicenter, randomized, double-blinded, placebo-controlled Phase 3 study of a microbiota suspension of intestinal microbes. Patients who have had at least one recurrence after a primary episode and have completed at least one round of standard-of-care oral antibiotic therapy or have had at least two episodes of severe Clostridioides difficile infection (CDI) resulting in hospitalization within the last year may be eligible for the study. Subjects who are deemed failures following the blinded treatment per the pre-specified treatment failure definition may elect to receive an unblinded dose of RBX2660.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blinded, placebo-controlled Phase 3 study of a microbiota suspension of intestinal microbes. The primary assessments for this study are (i) efficacy of RBX2660 as compared to a Placebo in preventing recurrent episodes of CDI and (ii) safety via assessment of adverse events. The primary efficacy analysis of the study will be a Bayesian hierarchical model, which formally incorporates data from a previous randomized Phase 2b study (Protocol 2014-01, NCT02299570) of RBX2660.

Follow-up office visits occur at weeks 1-, 4- and 8 after completing the blinded study treatment. Telephone assessments for adverse events occur during weeks 2, 3 and 6 after the study treatment and at months 3 and 6. Patients who have had at least one recurrence after a primary episode and have completed at least one round of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDI resulting in hospitalization within the last year may be eligible for the study. Study Subjects who are deemed failures following the blinded treatment per the pre-specified treatment failure definition may elect to receive an unblinded dose of RBX2660.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Medical record documentation of recurrent CDI per the study definition, that includes either: a) at least one recurrence after a primary episode and has completed at least one round of standard-of-care oral antibiotic therapy or b) has had at least two episodes of severe CDI resulting in hospitalization within the last year.
3. A positive stool test for the presence of toxigenic C. difficile within 30 days prior to or on the date of enrollment.
4. Is currently taking or was just prescribed antibiotics to control CDI related diarrhea at the time of enrollment.

[Note: Subject's CDI diarrhea must be controlled (<3 unformed/loose stools/day) while taking this course of antibiotics]

Exclusion Criteria:

1. Currently has continued CDI diarrhea despite being on antibiotics prescribed for CDI treatment.
2. Previous fecal transplant
3. History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis.
4. Diagnosis of irritable bowel syndrome (IBS) as determined by Rome III criteria.
5. Compromised immune system (e.g. immunosuppressed due to a medical condition or medication; current or recent (< 90 days) treatment with chemotherapy)
6. An absolute neutrophil count of <1000 cells/µL during screening.
7. Pregnant, breastfeeding, or intends to become pregnant during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teena Chopra, M.D., M.P.H., Study Chair — Wayne State University
Locations (63):
- United States (57):
  - Athens, Athens, Alabama
  - Dothan, Dothan, Alabama
  - Phoenix, Phoenix, Arizona
  - North Little Rock, North Little Rock, Arkansas
  - Lancaster, Lancaster, California
  - Los Angeles, Los Angeles, California
  - Oxnard, Oxnard, California
  - Sacramento, Sacramento, California
  - Aurora, Aurora, Colorado
  - Hamden, Hamden, Connecticut
  - Gainesville, Gainesville, Florida
  - Jacksonville, Jacksonville, Florida
  - Miami, Miami, Florida
  - Port Orange, Port Orange, Florida
  - Atlanta, Atlanta, Georgia
  - Idaho Falls, Idaho Falls, Idaho
  - Gurnee, Gurnee, Illinois
  - Highland Park, Highland Park, Illinois
  - Maywood, Maywood, Illinois
  - Lafayette, Lafayette, Indiana
  - Topeka, Topeka, Kansas
  - Wichita, Wichita, Kansas
  - Lexington, Lexington, Kentucky
  - New Orleans, New Orleans, Louisiana
  - Shreveport, Shreveport, Louisiana
  - Boston, Boston, Massachusetts
  - Detroit, Detroit, Michigan
  - Plymouth, Plymouth, Minnesota
  - Rochester, Rochester, Minnesota
  - St. Louis, St Louis, Missouri
  - Omaha, Omaha, Nebraska
  - Las Vegas, Las Vegas, Nevada
  - Teaneck, Teaneck, New Jersey
  - New York, New York, New York
  - North Massapequa, North Massapequa, New York
  - Rochester, Rochester, New York
  - Durham, Durham, North Carolina
  - Greenville, Greenville, North Carolina
  - Wilmington, Wilmington, North Carolina
  - Fargo, Fargo, North Dakota
  - Toledo, Toledo, Ohio
  - Portland, Portland, Oregon
  - Flourtown, Flourtown, Pennsylvania
  - Philadelphia, Philadelphia, Pennsylvania
  - Uniontown, Uniontown, Pennsylvania
  - Wyomissing, Wyomissing, Pennsylvania
  - Charleston, Charleston, South Carolina
  - Rapid City, Rapid City, South Dakota
  - Hixson, Hixson, Tennessee
  - Dallas, Dallas, Texas
  - Houston, Houston, Texas
  - West Jordan, West Jordan, Utah
  - Springfield, Springfield, Virginia
  - Winchester, Winchester, Virginia
  - Seattle, Seattle, Washington
  - Madison, Madison, Wisconsin
  - Marshfield, Marshfield, Wisconsin
- Canada (6):
  - Calgary, Calgary, Alberta
  - Edmonton, Edmonton, Alberta
  - Vancouver, Vancouver, British Columba
  - Victoria, Victoria, British Columbia
  - Fredericton, Fredericton, New Brunswick
  - Moncton, Moncton, New Brunswick

REFERENCES:
- [Background] Bakken JS. Feces transplantation for recurrent Clostridium difficile infection: US experience and recommendations. Microb Ecol Health Dis. 2015 May 29;26:27657. doi: 10.3402/mehd.v26.27657. eCollection 2015. No abstract available. PMID 26031677
- [Background] EISEMAN B, SILEN W, BASCOM GS, KAUVAR AJ. Fecal enema as an adjunct in the treatment of pseudomembranous enterocolitis. Surgery. 1958 Nov;44(5):854-9. No abstract available. PMID 13592638
- [Background] Miller MA, Louie T, Mullane K, Weiss K, Lentnek A, Golan Y, Kean Y, Sears P. Derivation and validation of a simple clinical bedside score (ATLAS) for Clostridium difficile infection which predicts response to therapy. BMC Infect Dis. 2013 Mar 25;13:148. doi: 10.1186/1471-2334-13-148. PMID 23530807
- [Derived] Lee C, Feuerstadt P, Louie T, Bancke L, Guthmueller B, Harvey A, Hoeyer F, Orenstein R, Dubberke ER, Khanna S. Integrated analysis of the safety of fecal microbiota, live-jslm in adults with recurrent Clostridioides difficile infection from five prospective clinical trials: an update. Therap Adv Gastroenterol. 2025 Nov 12;18:17562848251395566. doi: 10.1177/17562848251395566. eCollection 2025. PMID 41245385
- [Derived] Mishra R, Harvey A, Guo A, Tillotson G, Feuerstadt P, Khanna S, Shannon WD, Blount KF. Microbiome and metabolome changes after fecal microbiota, live-jslm, administration are associated with health-related quality of life improvements. Anaerobe. 2025 Dec;96:103006. doi: 10.1016/j.anaerobe.2025.103006. Epub 2025 Oct 18. PMID 41115624
- [Derived] Adamowicz E, Kraft CS, Ward T, Mehta N, Shannon WD, Mishra R, Blount KF. Decreased Antimicrobial Resistance Gene Richness Following Fecal Microbiota, Live-jslm (REBYOTA(R)) Administration: Post Hoc Analysis of PUNCH CD3. Open Forum Infect Dis. 2025 Jul 2;12(7):ofaf382. doi: 10.1093/ofid/ofaf382. eCollection 2025 Jul. PMID 40672762
- [Derived] Claypool J, Lindved G, Myers PN, Ward T, Nielsen HB, Blount KF. Microbiome compositional changes and clonal engraftment in a phase 3 trial of fecal microbiota, live-jslm for recurrent Clostridioides difficile infection. Gut Microbes. 2025 Dec;17(1):2520412. doi: 10.1080/19490976.2025.2520412. Epub 2025 Jun 24. PMID 40552763
- [Derived] Blount KF, Papazyan R, Ferdyan N, Srinivasan K, Gonzalez C, Shannon WD, Fuchs BC. Microbiome and Metabolome Restoration After Administration of Fecal Microbiota, Live-jslm (REBYOTA) for Preventing Recurrent Clostridioides difficile Infection. J Infect Dis. 2025 Jul 11;231(6):e1022-e1033. doi: 10.1093/infdis/jiae418. PMID 39172632
- [Derived] Feuerstadt P, Allegretti JR, Dubberke ER, Guo A, Harvey A, Yang M, Garcia-Horton V, Fillbrunn M, Tillotson G, Bancke LL, LaPlante K, Garey KW, Khanna S. Efficacy and Health-Related Quality of Life Impact of Fecal Microbiota, Live-jslm: A Post Hoc Analysis of PUNCH CD3 Patients at First Recurrence of Clostridioides difficile Infection. Infect Dis Ther. 2024 Jan;13(1):221-236. doi: 10.1007/s40121-023-00907-w. Epub 2024 Jan 18. PMID 38236515
- [Derived] Garey KW, Dubberke ER, Guo A, Harvey A, Yang M, Garcia-Horton V, Fillbrunn M, Wang H, Tillotson GS, Bancke LL, Feuerstadt P. Effect of Fecal Microbiota, Live-Jslm (REBYOTA [RBL]) on Health-Related Quality of Life in Patients With Recurrent Clostridioides difficile Infection: Results From the PUNCH CD3 Clinical Trial. Open Forum Infect Dis. 2023 Jul 20;10(8):ofad383. doi: 10.1093/ofid/ofad383. eCollection 2023 Aug. PMID 37564743
- [Derived] Khanna S, Assi M, Lee C, Yoho D, Louie T, Knapple W, Aguilar H, Garcia-Diaz J, Wang GP, Berry SM, Marion J, Su X, Braun T, Bancke L, Feuerstadt P. Efficacy and Safety of RBX2660 in PUNCH CD3, a Phase III, Randomized, Double-Blind, Placebo-Controlled Trial with a Bayesian Primary Analysis for the Prevention of Recurrent Clostridioides difficile Infection. Drugs. 2022 Oct;82(15):1527-1538. doi: 10.1007/s40265-022-01797-x. Epub 2022 Oct 26. PMID 36287379
- See also: Centers for Disease Control page last reviewed March 15, 2021; accessed March 01, 2022. — https://www.cdc.gov/healthcare-associated-infections/php/haic-eip/cdiff.html?CDC_AAref_Val=https://www.cdc.gov/hai/eip/cdiff-tracking.html
- See also: Sponsor website — http://www.rebiotix.com
- See also: Rebyota sponsor briefing book — https://www.fda.gov/advisory-committees/advisory-committee-calendar/vaccines-and-related-biological-products-advisory-committee-september-22-2022-meeting-announcement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from July 2017 to February 2020 at 44 medical clinics in the United States and Canada. Recruitment was performed by trained investigators and study coordinators.
Pre-assignment Details: A total of 320 subjects were enrolled (signed consent) of which 31 were screen failures.
  289 subjects were randomized: 193 to RBX2660 and 96 to placebo. Of the 289, 22 did not receive the allocated treatment.
  Therefore, a total of 267 subjects were randomized and treated: 180 subjects were treated with blinded RBX2660 treatment and 87 subjects were treated with blinded Placebo treatment.
Groups:
- Placebo: Placebo is normal saline administered rectally. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding
  Placebo: Placebo is normal saline solution administered rectally
- RBX2660: RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation United States Pharmacopeia (USP) solution and cryoprotectant
  RBX2660: RBX2660 is a microbiota suspension administered rectally
Period: Overall Study
Arm/Group | Placebo | RBX2660
Started | 87 | 180
Completed | 75 | 159
Not Completed | 12 | 21

BASELINE CHARACTERISTICS:
Groups:
- RBX2660: RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
  RBX2660: RBX2660 is a microbiota suspension administered rectally
- Total: Total of all reporting groups
Arm/Group | Placebo | RBX2660 | Total
Number analyzed (Participants) | 87 | 180 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 91 | 145
  >=65 years | 33 | 89 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (15.95) | 61.3 (16.81) | 60.1 (16.59)
Age, Continuous [Median (Full Range); unit: years] | 60.0 [26 to 86] | 64.0 [19 to 93] | 63.0 [19 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 123 | 183
  Male | 27 | 57 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 80 | 168 | 248
  Unknown or Not Reported | 3 | 10 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 78 | 168 | 246
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 51 | 77
  United States | 61 | 129 | 190
Clostridioides difficile infection (CDI) History [Count of Participants; unit: Participants] — Number of CDI Episodes before Blinded Treatment
  Participants
    <=3 | 59 | 111 | 170
    >3 | 28 | 69 | 97
Antibiotic Screening [Count of Participants; unit: Participants] — Antibiotics taken for qualifying CDI event prior to Blinded Treatment
  Participants
    Vancomycin alone | 78 | 157 | 235
    Vancomycin in combination | 2 | 5 | 7
    Fidaxomicin | 5 | 12 | 17
    Other | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of RBX2660 Compared to Placebo Through 8 Weeks
Description: The primary efficacy endpoint was the absence of CDI diarrhea for 8 weeks after study treatment. The model-estimated rate of treatment success, that is the model-estimated percentage of participants that met the primary efficacy endpoint, was estimated using a Bayesian hierarchical model, which formally incorporated data from a previous randomized Phase 2B study (NCT02299570) of RBX2660.
Time Frame: 8 weeks after completing the study treatment
Population: The modified Intent-To-Treat (mITT) Population included all randomized patients who successfully received blinded treatment, excluding those who discontinued from the study for reasons not related to CDI symptoms prior to evaluation of Treatment Success for the primary endpoint.
Measure: Number (95% Confidence Interval); unit: Model-estimated percent of participants
Arm/Group | Placebo | RBX2660
Number analyzed (Participants) | 85 | 177
Model-estimated percent of participants | 57.5 [48.1 to 67.1] | 70.6 [64.1 to 76.8]
Statistical Analysis 1: Comparison: Placebo vs RBX2660; A hierarchical, closed-testing procedure (Bayesian hierarchical model) was utilized for the primary endpoint. The Bayesian hierarchical model formally incorporated data from the previous Phase 2B study (NCT02299570) of RBX2660. This analysis tested the hypothesis that the response rate of RBX2660 was superior to Placebo and was performed at the nominal 0.00125 and 0.025 one-sided levels; Test type: Superiority; Treatment Difference = 13.1, 95% CI 2-sided [2.3 to 24.0] — The Bayesian posterior probability of superiority was 0.99136. This value exceeded the pre-specified threshold of 0.9750338 (nominal 0.025 one-sided level)

2. Secondary Outcome: Sustained Clinical Response Through 6 Months After Blinded Treatment
Description: The rates of Sustained Clinical Response (i.e., the occurrence of new CDI infections from baseline through 6 months) was assessed by either the rate of new CDI infections after treatment success at 8 weeks (durability) or the frequency of total CDI infections from baseline through 6 months.
  Sustained Clinical Response was compared between the RBX2660 group and the control group using a chi-square test. Patients who exited prior to their 6-month follow-up were conservatively counted as a Treatment Failure
Time Frame: 6 months after completing the study treatment
Population: The mITT population included all randomized patients who successfully received blinded treatment, excluding those who discontinued from the study for reasons not related to CDI symptoms prior to evaluation of Treatment Success for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RBX2660
Number analyzed (Participants) | 85 | 177
Participants
  From 8 weeks through 6 months (Durability): number analyzed (Participants) | 53 | 126
  From 8 weeks through 6 months (Durability) | 48 | 116
  Through 6 months | 48 | 116
Statistical Analysis 1: Comparison: Placebo vs RBX2660; Test type: Superiority; p = 0.156, Chi-squared — P-value for secondary outcome evaluated from baseline through 6 months

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from enrollment through 6 months after the last dose received, which may have been blinded placebo, blinded RBX2660 or an open label dose of RBX2660.
Description: Treatment emergent adverse events, defined as adverse events occurring after exposure to the study drug (placebo or RBX2660) are presented. Participants were systematically asked about any occurrences of adverse events at each contact point (in office or scheduled phone call) and via a daily diary for one week after each dose.
Groups:
- Placebo Only: Placebo randomized subjects who did not receive an unblinded RBX2660.
  Placebo is normal saline administered rectally. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding
  Placebo: Placebo is normal saline solution administered rectally
- RBX2660 Only: RBX2660 randomized subjects who did not receive an unblinded RBX2660.
  RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
  RBX2660: RBX2660 is a microbiota suspension administered rectally
- Blinded Placebo/Open-label RBX2660 (Blinded Period): Placebo randomized subjects who went on to receive an unblinded RBX2660 (blinded period).
  Treatment-emergent adverse events (TEAEs) are defined as any adverse events occurring on or after the blinded treatment. For TEAEs counted in open-label treatment period, TEAEs are reported with an onset date on or after the date of the open-label treatment through 6 months timeframe.
  Placebo is normal saline rectally administered. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding.
  RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
- Blinded RBX2660/Open-label RBX2660 (Blinded Period): RBX2660 randomized subjects who went on to receive an unblinded RBX2660 (blinded period).
  Treatment-emergent adverse events (TEAEs) are defined as any adverse events occurring on or after the blinded treatment. For TEAEs counted in open-label treatment period, TEAEs are reported with an onset date on or after the date of the open-label treatment through 6 months timeframe.
  Placebo is normal saline rectally administered. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding.
  RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
- Blinded Placebo/Open-label RBX2660 (Open-label Period): Placebo randomized subjects who went on to receive an unblinded RBX2660 (open-label period).
  Treatment-emergent adverse events (TEAEs) are defined as any adverse events occurring on or after the blinded treatment. For TEAEs counted in open-label treatment period, TEAEs are reported with an onset date on or after the date of the open-label treatment through 6 months timeframe.
  Placebo is normal saline rectally administered. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding.
  RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
- Blinded RBX2660/Open-label RBX2660 (Open-label Period): RBX2660 randomized subjects who went on to receive an unblinded RBX2660 (open-label period).
  Treatment-emergent adverse events (TEAEs) are defined as any adverse events occurring on or after the blinded treatment. For TEAEs counted in open-label treatment period, TEAEs are reported with an onset date on or after the date of the open-label treatment through 6 months timeframe.
  Placebo is normal saline rectally administered. Packaging and labeling are identical to the packaging and labeling for RBX2660 to support the study blinding.
  RBX2660 is a rectally administered microbiota suspension in a 0.9% sodium chloride irrigation USP solution and cryoprotectant
Arm/Group | Placebo Only | RBX2660 Only | Blinded Placebo/Open-label RBX2660 (Blinded Period) | Blinded RBX2660/Open-label RBX2660 (Blinded Period) | Blinded Placebo/Open-label RBX2660 (Open-label Period) | Blinded RBX2660/Open-label RBX2660 (Open-label Period)
All-Cause Mortality (participants affected / at risk) | 0/63 | 1/139 | 0/24 | 0/41 | 0/24 | 1/41
Serious Adverse Events (participants affected / at risk) | 5/63 | 9/139 | 1/24 | 3/41 | 1/24 | 5/41
Other Adverse Events (participants affected / at risk) | 23/63 | 56/139 | 5/24 | 3/41 | 10/24 | 19/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Only (N=63) | RBX2660 Only (N=139) | Blinded Placebo/Open-label RBX2660 (Blinded Period) (N=24) | Blinded RBX2660/Open-label RBX2660 (Blinded Period) (N=41) | Blinded Placebo/Open-label RBX2660 (Open-label Period) (N=24) | Blinded RBX2660/Open-label RBX2660 (Open-label Period) (N=41)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multimorbidity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Only (N=63) | RBX2660 Only (N=139) | Blinded Placebo/Open-label RBX2660 (Blinded Period) (N=24) | Blinded RBX2660/Open-label RBX2660 (Blinded Period) (N=41) | Blinded Placebo/Open-label RBX2660 (Open-label Period) (N=24) | Blinded RBX2660/Open-label RBX2660 (Open-label Period) (N=41)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 8 (11) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 24 (27) | 4 (4) | 1 (2) | 2 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 28 (40) | 2 (2) | 1 (2) | 5 (5) | 9 (12)
Flatulence (Gastrointestinal disorders) | 0 (0) | 8 (10) | 1 (3) | 1 (3) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 14 (15) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (3) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT03244644/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03244644/SAP_001.pdf